CLINICAL TRIAL: NCT05661253
Title: Ultrasound Guided Modified Versus Conventional Serratus Anterior Plane Block as a Preemptive Analgesia for Unilateral Video-Assisted Thoracoscopic Surgery
Brief Title: Modified Versus Conventional Serratus Anterior Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba M Fathi, prof/Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZU-IRB # 10061
Record Dates: First submitted 2022-12-01; First posted 2022-12-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): will take general anesthesia without nerve block
- SAP block group (Active Comparator): After sterilization of the skin and draping, the high frequency linear probe of Sonosite M Turbo ultrasonography (FUJIFIM sonosite, Inc., Bothell, WA, USA) will be placed at the level of the midclavicular line in a sagittal plane. The second rib will be recognized at the axillary artery. The probe will be moved downward to count the ribs until the level of the ﬁfth rib in the mid-axillary line. At this time, the latissimus dorsi muscle (lying superficial) and the serratus anterior muscle (lying deep) will be clearly visualized under ultrasound . Next, A 22-gauge, 80 mm needle (Stimuplex D, B-Braun, Germany) will be inserted in plane relative to the ultrasound probe between the latissimus dorsi and the serratus anterior muscle. After confirming negative aspiration of blood, 1 ml normal saline will be injected for hydro-dissection sign to verify the needle tip, then a volume of 25 ml 0.25% bupivacaine will be injected superficially to serratus anterior muscle. .
  Interventions: Drug: 25 ml of bupivacaine 0.25% via serratus anterior block
- modified SAP block group (Active Comparator): The patient will be placed in the lateral decubitus position according to the selected site of surgical intervention. After sterilization of the skin and draping, the high frequency linear probe of Sonosite M Turbo ultrasonography ( FUJIFIM sonosite, Inc., Bothell, WA, USA) will be placed horizontally midway between tip of the scapula and posterior axillary line to identify the view of latissimus dorsi(lying superficial) and serratus anterior muscle(lying deep) over either the sixth or seventh rib. A 22-gauge, 80 mm needle (Stimuplex D, B-Braun, Germany) will be inserted in plane relative to the ultrasound probe from posteromedial to anterolateral direction toward posterior axillary line till reaching the interfacial plane between latissimus dorsi and serratus anterior muscle . After confirming negative aspiration of blood, 1 ml normal saline will be injected for hydro-dissection sign to verify the needle tip, then a volume of 25 ml 0.25% bupivacaine will be injected .
  Interventions: Drug: 25 ml of bupivacaine 0.25% via modified serratus anterior palne block

INTERVENTIONS:
Drug: 25 ml of bupivacaine 0.25% via serratus anterior block — patients will receive conventional serratus anterior plane block with a volume of 25 ml of bupivacaine 0.25% followed by induction of general anesthesia,
  Arms: SAP block group
Drug: 25 ml of bupivacaine 0.25% via modified serratus anterior palne block — patients will receive modified serratus anterior plane block with a volume of 25 ml of bupivacaine 0.25% followed by induction of general anesthesia.
  Arms: modified SAP block group

SUMMARY:
comparing preemptive analgesia with ultrasound guided modified serratus anterior plane block versus ultrasound guided serratus anterior plane block

DETAILED DESCRIPTION:
comparing the quality of postoperative analgesia and opioid consumption in patients undergoing Video-Assisted Thoracoscopic Surgery when using preemptive analgesia with ultrasound guided modified serratus anterior plane block versus ultrasound guided serratus anterior plane block

ELIGIBILITY:
Inclusion Criteria:

* Patient consent.
* both sex.
* Age: 21-70 years old.
* BMI: 18- 30 kg/m2
* ASA: I and II.
* Scheduled for elective unilateral Video-Assisted thoracoscopy under general anesthesia.

Exclusion Criteria:

* History of allergy to the local anesthesia agents used in this study,
* Skin lesion at needle insertion site,
* Those receiving anticoagulant therapy or having bleeding disorders
* Patients with history of chronic pain and taking analgesics,
* Patients with sepsis and Significant cardiac, liver or renal diseases
* Uncooperative patients or with psychiatric disorders.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
tramadol consumption | at 24 hours postoperative
  The amount of tramadol consumption at 24

SECONDARY OUTCOMES:
Time of performance | from ultrasound probe positioning till the end of the block procedure
  Time of performance of block defined as time from ultrasound probe positioning till the end of the block procedure
Time to first dose of rescue analgesia | during the first postoperative 24 hours
  Time to first dose of rescue analgesia (VAS > 3) after surgery
Patient satisfaction | at 24 hous post operative
  Patient satisfaction with analgesia in the first 24hours postoperative hours will be Likert scale where 5 is very satisfied and 0 is very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Fathi, Principal Investigator — faculty of human medicine ,zagazig university
Locations (1):
- Heba M Fathi, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abd Ellatif SE, Galal Eldin AM, Ali ES, Fathi HM. Ultrasound-guided modified versus conventional serratus anterior plane block as a preemptive analgesic for unilateral video-assisted thoracoscopic surgery. BMC Anesthesiol. 2025 Aug 29;25(1):435. doi: 10.1186/s12871-025-03314-5. PMID 40883665